CLINICAL TRIAL: NCT02412956
Title: Quit4Baby: Reaching Pregnant Smokers With Health Information Via Text
Brief Title: SmokefreeMOM: Reaching Pregnant Smokers With Health Information Via Text Messaging
Acronym: SmokefreeMOM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: George Washington University (Other)
Responsible Party: Principal Investigator, Lorien Abroms, Associate Professor, George Washington University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R15CA167586 (NIH)
Record Dates: First submitted 2015-03-31; First posted 2015-04-09 (Estimated); Results first posted 2021-11-26 (Actual); Last update posted 2021-11-26 (Actual); Status verified 2021-10

CONDITIONS: Pregnancy; Smoking Cessation
Keywords: mHealth
MeSH Terms: conditions — Smoking Cessation

ARMS (3):
- Control (No Intervention): pamphlet
- Intervention (text) (Experimental): SmokefreeMOM text messaging program
  Interventions: Behavioral: SmokefreeMOM Text
- Intervention Plus (text+quitline) (Experimental): SmokefreeMOM text messaging program + state quitline
  Interventions: Behavioral: SmokefreeMOM Text

INTERVENTIONS:
Behavioral: SmokefreeMOM Text
  Arms: Intervention (text); Intervention Plus (text+quitline)

SUMMARY:
Despite the great health benefits associated with smoking cessation in pregnancy to both mother and baby, few studies to date have examined the applications of text messaging or other communication technologies for smoking cessation in this population. This project is the first step in developing a new dissemination strategy for reaching pregnant smokers. This research will explore how a state-of -the-art, interactive and intensive, text messaging program, SmokefreeMoms Text, can promote smoking cessation in pregnant smokers. This program may have the potential to reach pregnant smokers who are not currently being reached with traditional smoking cessation services. The study Aims are: 1) to elicit qualitative feedback from pregnant smokers and recent quitters (in the past month) about the concept of SmokefreeMoms, the proposed message protocols in SmokefreeMoms, and the proposed messages in SmokefreeMoms (Phase 1); 2) To develop and pilot test a prototype of SmokefreeMoms which is consistent with Clinical Practice Guidelines (Phase 2), and 3) To conduct a formative evaluation of SmokefreeMoms 1.0 with pregnant smokers and recent quitters (Phase 3). 4) To measure the likelihood that pregnant women who smoke cigarettes will join an SMS program by responding to different types of recruitment messages.

ELIGIBILITY:
Inclusion Criteria:

1. pregnant,
2. smoke or quit in the past 2 weeks,
3. has a data plan or an unlimited text messaging plan on her cell in order to avoid charges for texts,
4. an English speaker.

Exclusion Criteria:

1. not pregnant
2. not currently smoking (or within past 2 weeks)
3. not able to receive text messages
4. not an English speaker

Ages: 13 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 99 (Actual)
Dates: Start 2013-01; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Medstar Hospital, Washington D.C., District of Columbia, United States

REFERENCES:
- [Derived] Palmer MJ, Henschke N, Bergman H, Villanueva G, Maayan N, Tamrat T, Mehl GL, Glenton C, Lewin S, Fonhus MS, Free C. Targeted client communication via mobile devices for improving maternal, neonatal, and child health. Cochrane Database Syst Rev. 2020 Jul 14;8(8):CD013679. doi: 10.1002/14651858.CD013679. PMID 32813276
- [Derived] Abroms LC, Chiang S, Macherelli L, Leavitt L, Montgomery M. Assessing the National Cancer Institute's SmokefreeMOM Text-Messaging Program for Pregnant Smokers: Pilot Randomized Trial. J Med Internet Res. 2017 Oct 3;19(10):e333. doi: 10.2196/jmir.8411. PMID 28974483

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 11 obstetrics-gynecology clinics from 9/5/14 to 5/25/16; 9 from Medstar Health, one GWU MFA, and the other Capital Women's Care. The recruitment occurred via the electronic medical record as smokers and pregnant and sent a letter about the study. Subjects were recruited by physicians at the time of visit and were called by study staff.
Groups:
- Intervention (Text): SmokefreeMOM text messaging program
  SmokefreeMOM Text
- Intervention Plus (Text+Quitline): SmokefreeMOM text messaging program + state quitline
  SmokefreeMOM Text
Period: Overall Study
Arm/Group | Control | Intervention (Text) | Intervention Plus (Text+Quitline)
Started | 44 | 47 | 8
Completed | 35 | 30 | 8
Not Completed | 9 | 17 | 0

BASELINE CHARACTERISTICS:
Population: As very few participants in the SmokefreeMOM + Quitline group reported receiving quitline services (n=2) and because the group was small, a decision was made to combine the SmokefreeMOM + Quitline group (n=8) with the SmokefreeMOM group (n=47) and to compare these combined groups (referred to as "the intervention group") to the control group (n=44). Before combining groups, baseline demographic characteristics between these 2 groups were compared with no major differences observed.
Groups:
- Intervention: SmokefreeMOM text messaging program and SmokefreeMOM text messaging program+ Quitline
- Total: Total of all reporting groups
Arm/Group | Control | Intervention | Total
Number analyzed (Participants) | 44 | 55 | 99
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 44 | 55 | 99
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.25 (4.78) | 27.18 (4.98) | 27.66 (4.90)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 55 | 99
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 44 | 55 | 99

OUTCOME MEASURES:

1. Primary Outcome: Smoking Abstinence
Description: 7-day point prevalence abstinence measured by Self-Report and Confirmed with Saliva Cotinine
Time Frame: 3 months
Measure: Number; unit: participants
Groups:
- Intervention: SmokefreeMOM text messaging program and SmokefreeMOM text messaging program + state quitline
Arm/Group | Control | Intervention
Number analyzed (Participants) | 44 | 55
participants | 4 | 8

ADVERSE EVENTS:
Arm/Group | Control | Intervention
All-Cause Mortality (participants affected / at risk) | 0/44 | 0/55
Serious Adverse Events (participants affected / at risk) | 0/44 | 0/55
Other Adverse Events (participants affected / at risk) | 0/44 | 0/55

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No